CLINICAL TRIAL: NCT06992297
Title: Clinical Evaluation of Long-term Sequelae in Patients With Severe Plasmodium Falciparum Malaria
Acronym: SMAEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AP-HM; 2025-A00117-48 (Other: IDRCB)
Record Dates: First submitted 2025-05-19; First posted 2025-05-28 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-09

CONDITIONS: Falciparum Malaria
MeSH Terms: conditions — Malaria, Falciparum | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- malaria patient (Other)
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — a standardised, structured questionnaire, validated by the department's clinicians, to assess the physical, cognitive and psychological after-effects.

SUMMARY:
Malaria, endemic in 85 countries, remains a major concern. By 2022, there will be 249 million cases and 608,000 deaths, 94% of them in Africa. In France, 4995 cases of imported malaria were reported in 2021, with 15% of severe forms and a fatality rate of 2.5%. Long-term sequelae, such as kidney failure and neurological disorders, are well documented in children, but few studies have focused on adults.

the main objective is to describe and estimate the frequency of long-term sequelae of severe imported malaria treated at our centre.

the aim is to compare long-term neurological sequelae between neuromalaria and severe malaria without neurological disorders. In addition, the investigator aim to identify the clinical, radiological and biological factors associated with sequelae in order to improve post-hospitalisation follow-up. Finally, the investigator aim to describe acute complications arising at diagnosis and during hospitalisation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years of age
* Have been diagnosed with severe malaria according to WHO criteria and have been treated between 1/1/2018 and 321/12/2024 at the AP-HM
* Have been treated with Artesunate IV (MALACEF®) (at least one dose)
* Patient who has received information about the study and has not expressed opposition
* Patient benefiting or entitled to benefit from a social security scheme

Exclusion Criteria:

* Patients with advanced neurodegenerative pathology pre-existing the malaria attack
* Subjects covered by articles L1121-5 to 1121-8 of the Public Health Code (minor patients, patients of legal age under guardianship, curatorship or safeguard of justice, patients deprived of their liberty, pregnant or breast-feeding women),
* Persons who do not understand French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2025-06-17 (Actual); Primary Completion 2025-09-13 (Actual); Study Completion 2025-09-13 (Actual)

PRIMARY OUTCOMES:
frequency of long-term sequelae of severe malaria | 12 months
  Assessment of after-effects one year after diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Francois CREMIEUX, Study Director — APHM; Coralie L'OLLIVIER, doctor, Principal Investigator — APHM
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France